CLINICAL TRIAL: NCT00409318
Title: Effects of TNF-Alpha Antagonism in Patients With the Metabolic Syndrome (I)
Brief Title: Study of TNF-Antagonism in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Steven Grinspoon, M.D., MGH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-P-001699
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Metabolic Syndrome
Keywords: Inflammation; Visceral adiposity; TNF; CRP; Adiponectin; Insulin resistance; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Insulin Resistance | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Etanercept
  Interventions: Drug: Etanercept
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — 50 mg SC q week
  Other Names: Enbrel
  Arms: 1
Drug: Placebo — SC q week
  Arms: 2

SUMMARY:
This study investigates whether blockade of TNF will result in reduced inflammatory indices in patients with the metabolic syndrome

DETAILED DESCRIPTION:
Metabolic syndrome is an increasingly prevalent disorder associated with elevated risks of type II DM (diabetes mellitus) and cardiovascular morbidity and mortality. A subclinical inflammatory state is thought to contribute to the pathophysiology of metabolic syndrome, insulin resistance, and coronary artery disease (CAD). TNF-alpha is an inflammatory cytokine that is increased in a spectrum of inflammatory diseases as well as in insulin resistance. TNF-alpha antagonists are clinically effective in the inflammation of arthritides, but have not been examined in the metabolic syndrome population. Moreover, data suggests that adiponectin, a recently discovered adipocytokine that may protect against the development of insulin resistance and atherosclerosis, may be downregulated by TNF-alpha. We propose a study in which we administer etanercept, a TNF-alpha receptor fusion protein, to subjects with metabolic syndrome to examine its effect on inflammatory markers,CRP, adiponectin and insulin resistance. This would be the first study to investigate the anti-inflammatory properties and insulin sensitizing potential of TNF-alpha blockade on the growing population with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria based on a modified WHO definition of metabolic syndrome

1. Hyperinsulinemia in the upper quartile of the non-diabetic population defined as >= 10 mU/mL (Framingham Data, oral communication,James Meigs, MD) or fasting glucose 110-126 mg/dL

   Plus two of the following:
2. Abdominal obesity defined by waist hip ratio > 0.90 for men and > 0.85 for women or BMI > 30 kg/m2
3. Dyslipidemia including serum triglycerides ³ 150 mg/dl or serum HDL < 0.9 mmol/L for men (35 mg/dL) and < 1.0 mmol/L (39mg/dL) for women
4. Hypertension defined as blood pressure >= 140/90 or on medication

Exclusion Criteria:

1. Positive PPD (³ 5mm induration) on screening
2. Current Infection
3. Therapy with glucocorticoid or immunosuppressant at time of recruitment or within past 3 months
4. Reception of live vaccine within 1 week of recruitment
5. History of blood dyscrasia including any kind of anemia, thrombocytopenia, pancytopenia. Women with a reversible cause of anemia that has resolved will be eligible.
6. History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers who will be eligible)
7. History of organ transplantation
8. History of CNS demyelinating disorder or any first degree relative with multiple sclerosis
9. History of CHF classes I-IV
10. Current use of insulin, any oral anti-hyperglycemic agents, pentoxyfylline, beta-agonists
11. Current use of fibrate or niacin
12. Initiation of statin therapy within prior 6 weeks or expecting a change in statin dose over the upcoming 3 months
13. Hemoglobin < 11 g/dl
14. Positive pregnancy test
15. Women of child-bearing potential not currently using non-hormonal birth control methods including barrier methods (IUD, condoms, diaphragms) or abstinence
16. Patients with known autoimmune or inflammatory conditions (excluding patients with stable, treated hypothyroidism)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2004-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
CRP | 4 weeks

SECONDARY OUTCOMES:
Insulin resistance | 4 weeks
Muscle adiposity | 4 weeks
High molecular weight adiponectin | 4 weeks
resistin | 4 weeks
leptin | 4 weeks
TNF-R1 | 4 weeks
TNF-R2 | 4 weeks
weight | 4 weeks
WBC | 4 weeks
Lipids | 4 weeks
IL-6 | 4 weeks
Fibrinogen | 4 weeks
adiponectin | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, Principal Investigator — MGH
Locations (1):
- MGH, Boston, Massachusetts, United States

REFERENCES:
- [Result] Bernstein LE, Berry J, Kim S, Canavan B, Grinspoon SK. Effects of etanercept in patients with the metabolic syndrome. Arch Intern Med. 2006 Apr 24;166(8):902-8. doi: 10.1001/archinte.166.8.902. PMID 16636217
- [Derived] Zanni MV, Stanley TL, Makimura H, Chen CY, Grinspoon SK. Effects of TNF-alpha antagonism on E-selectin in obese subjects with metabolic dysregulation. Clin Endocrinol (Oxf). 2010 Jul;73(1):48-54. doi: 10.1111/j.1365-2265.2009.03741.x. PMID 19878508